CLINICAL TRIAL: NCT03605290
Title: Comparison Between Two Operational Techniques for Total Knee Replacement: A Prospective, Case Control, Double Blinded Study
Brief Title: Comparison Between Two Operational Techniques for Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Uriel Giwnewer, Principal investigator, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 003418EMC
Record Dates: First submitted 2018-06-18; First posted 2018-07-30 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Gait, Unsteady; Knee Arthropathy; Surgery
Keywords: total knee replacement; gait analysis; PROMS; mechanical aligment; kinematic alignment
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The operative technique (Kinematic Vs. Mechanically aligned) is not revealed to the patient, investigator and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanically aligned TKR (Active Comparator): patients were operated using the standard mechanically aligned technique
  Interventions: Diagnostic Test: REHAGAIT ANYLIZER
- Kinematically aligned TKR (Experimental): patients were operated using the newer mechanically aligned technique
  Interventions: Diagnostic Test: REHAGAIT ANYLIZER

INTERVENTIONS:
Diagnostic Test: REHAGAIT ANYLIZER — Gait analysis instrumentation

SUMMARY:
Advance Knee osteoarthritis is treated by Total knee replacement. Since the first TKR in 1973 there has been continuous advance in implant technology as well as operative technique, yet current patient satisfaction after the procedure is accepted to be about 80%.

There are a few operative techniques to perform TKR. Until recently the most common technique is the anterior approach to the knee and then using mechanical instrumentation to make the bone cuts for the femur and tibia. A second popular technique is the anterior approach to the knee and then using a kinematic alignment to make the bone cuts.

The investigators wish to compare short term results of the two operative techniques as evidenced in patient objective functional scores and also by evaluating the gait of the patients by using the REHAGAIT ANALYZER PRO by HASOMED inc. Magdeburg Germany.

ELIGIBILITY:
Inclusion Criteria:

- Patients after total knee replacement which was performed in our ward.

Exclusion Criteria:

* Less than 6 months have passed after the procedure
* Inability to understand and fill out PROMS questionnaires.
* Inability to walk without aids for at least 20 meters.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
PROMS | At least 6 months post operatively
  The patients will fill out functionala and quality of life assessment questionnaires
Gait analysis | At least 6 months post operatively
  The patients will perform a gait analysis using the REHAGAIT system.

CONTACTS AND LOCATIONS:
Locations (1):
- haemek MC, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided